CLINICAL TRIAL: NCT06964230
Title: A Phase 2b/3 Randomized, Double-Blind, Placebo-Controlled Multi-Center Study to Evaluate the Safety and Efficacy of T3D-959 in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: A Phase 2b/3 Clinical Study Evaluating T3D-959 in Mild-to-Moderate Alzheimer's Disease Subjects
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: T3D Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, John Didsbury, Chief Executive Officer, T3D Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T3D959-301
Record Dates: First submitted 2025-04-14; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
Keywords: T3D-959; Mild-to-Moderate Alzheimer's Disease Severity; New Drug Treatment Being Tested; Once-a-day oral drug administration; Phase 2b/3 Study T3D959-301; Brain Metabolism
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo, matching T3D-959 active capsules (Placebo Comparator): Placebo Comparator: Placebo, matching T3D-959 active capsules, is pregelatinized starch NF, magnesium stearate NF, and size 0, hard gelatin, white/white, opaque, unmarked capsules. Subjects randomized to placebo will ingest two size 0 placebo capsules once per day in the morning.
  Interventions: Other: Placebo Comparator
- 30mg T3D-959 (Experimental): Experimental: 30mg T3D-959 Arm Description: Experimental: T3D-959 30 mg dose: T3D-959 is a small molecule dual nuclear receptor agonist that regulates transcription of genes, in particular those involved in glucose energy and lipid metabolism. T3D-959 is 15-times more potent for PPAR delta than for the secondary target of the drug, PPAR gamma. The 15 mg strength contains 15mg T3D-959, pregelatinized starch NF, magnesium stearate NF, and size 0, hard gelatin, white/white, opaque, unmarked capsules. Subjects will ingest two size 0, 15mg capsules once per day in the morning.
  Interventions: Drug: T3D-959

INTERVENTIONS:
Drug: T3D-959 — Experimental:
  T3D-959 30 mg dose: T3D-959 is a small molecule dual nuclear receptor agonist that regulates transcription of genes, in particular those involved in glucose energy and lipid metabolism. T3D-959 is 15-times more potent for PPAR delta than for the secondary target of the drug, PPAR gamma. The 15 mg strength capsules contain 15mg T3D-959, pregelatinized starch NF, magnesium stearate NF, and size 0, hard gelatin, white/white, opaque, unmarked capsules. Subjects will ingest two size 0, 15mg capsules once per day in the morning.
  Arms: 30mg T3D-959
Other: Placebo Comparator — Placebo used to compare to T3D-959 drug
  Arms: Placebo, matching T3D-959 active capsules

SUMMARY:
This study is a Phase 2b/3 clinical trial of a new candidate drug (T3D-959) to treat patients with mild-to-moderate Alzheimer's. The aims of the trial are to affirm potential therapeutic efficacy and safety observed in earlier clinical trials and assess the potential to modify the course of disease. The drug will be compared to placebo and administered orally to patients once a day for 78 weeks.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled study of T3D-959 30mg in subjects with clinical mild-to-moderate Alzheimer's Disease and a biological diagnosis of AD pathology, as defined by a validated plasma biomarker (presently %p-tau217 plasma biomarker). This study is designed as a seamless group sequential design where estimates of treatment effect on cognitive and functional scales will be evaluated in an interim analysis by independent statisticians. The sample size will be re-estimated to ensure the study is sufficiently powered to demonstrate efficacy of T3D-959 in cognition and function.

Subjects will be assigned to one of two treatment arms (1:1 ratio) in a randomized, double-blind fashion, stratified by sex and ApoE4 genotype. Study medication will be taken once daily for 78 weeks. Safety/tolerability, efficacy and exploratory assessments will be evaluated for changes from baseline to end of treatment (78 weeks). Subjects will be followed for four weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged 50-90 years old inclusive at the time of Informed Consent
2. Subject (or legal representative) and caregiver must sign an Informed Consent to participate in the study.
3. Subject has a caregiver, an identified adult who, in the opinion of the investigator, has sufficient contact to knowledgeably report on the subject's cognition, function, behavior, safety, compliance and adherence. Same caregiver should, whenever possible, assist the subject throughout the duration of the trial
4. Subject has a biological diagnosis of AD pathology, as assessed by a validated plasma biomarker (presently %p-tau217 plasma biomarker), according to the NIA-AA (National Institute of Aging - Alzheimer's Association) criteria at screening
5. Subject has a clinical diagnosis of mild to moderate AD (Stage 4 or 5) according to the NIA-AA (National Institute of Aging - Alzheimer's Association) criteria at screening
6. Meets criteria for mild-to-moderate cognitive impairment with Mini-Mental State Examination (MMSE) score of 14 through 26 at the screening visit.
7. Modified Hachinski < 4 at screening
8. Clinical Dementia Rating is 0.5 to 2.0 at screening
9. Visual and auditory acuity adequate for neuropsychological testing
10. Medical stability for this study as confirmed by review of records, comprehensive physical exam, neurological exam, and laboratory tests
11. Washout and stability of all concurrent medication according to the exclusion criteria listed below
12. Able to swallow oral medications

Exclusion Criteria:

1. Subject has a current diagnosis of a significant psychiatric illness per the Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) including but not limited to major depressive disorder, anxiety disorders and is in an acute phase/episode; or the subject has a current diagnosis or history of schizophrenia or bipolar disorder; or has current signs of suicidality or history of suicide attempt
2. Subject with untreated clinical depression at screening; Geriatric Depression Scale (GDS) Short Form > 9
3. Evidence of clinically significant lesion(s) on brain MRI at Screening that could indicate a dementia diagnosis other than Alzheimer's disease
4. Other significant pathological findings on brain MRI at screening, including but not limited to: more than 4 microhemorrhages (defined as 10 millimeter [mm] or less at the greatest diameter); a single macrohemorrhage >10 mm at greatest diameter; an area of superficial siderosis; evidence of vasogenic edema; evidence of cerebral contusion, encephalomalacia, aneurysms, vascular malformations, or infective lesions; evidence of multiple lacunar infarcts or stroke involving a major vascular territory, severe small vessel, or white matter disease; space occupying lesions; or brain tumors (however, lesions diagnosed as meningiomas or arachnoid cysts and <1 centimeter [cm] at their greatest diameter need not be exclusionary)
5. Subject has a current diagnosis of a neurological disease other than AD, which has or could result in cognitive impairment, including, but not limited to, any of the following:

   1. History of clinically significant stroke or multiple strokes as ascertained by history and/or brain imaging findings, or history of TIA's within 12 months prior to baseline
   2. History of serious brain infection
   3. History of or current space occupying cerebral lesion
   4. History of clinically significant concussion or repeated head trauma associated with sustained cognitive impairment in the last 5 years
   5. Huntington's Disease
   6. Parkinson's Disease
   7. Dementia predominantly of a non-Alzheimer's type (vascular dementia, frontotemporal dementia, Parkinson's dementia, substance-induced dementia)
   8. Normal pressure hydrocephalus
   9. History of seizures (except for childhood febrile) or epilepsy
6. With glycosylated hemoglobin (HbA1c) ≥ 10 at screening
7. Subject with a diagnosis of unstable diabetes
8. Subject with clinically significant thyroid disease at screening TSH >5 and abnormal T3/T4
9. Subject has any evidence of hepatic impairment or renal insufficiency, including any of the following values at the screening visit:

   1. Serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) value that is twice the upper limit of normal
   2. A serum total bilirubin value that exceeds 2 mg/dL
   3. Serum creatinine level >1.5 mg/dL in men or > 1.4 mg/dL in women
   4. Positive urinalysis consistent with renal impairment
   5. Estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2
   6. Gamma glutamyl-transpeptidase (GGT) twice the upper limit of normal
10. Subject is positive for hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (HCV) antibodies at the screening visit
11. Subject has a history of moderate or severe congestive heart failure, NYHA class III or IV, within 12 months prior to baseline
12. Subject has experienced a previous cardiovascular event (myocardial infarct, by-pass surgery, or PTCA) within the past 6 months prior to the baseline (visit 2)
13. Subject has blood pressure reading at screening that is greater than 160/100 mmHg. Subjects with elevated BP will be allowed at the discretion of the principal investigator. Blood pressure will be measured after the subject has been supine for at least 5 minutes followed by repeat measurement after standing for at least 3 minutes. Subjects will be excluded if a significant diastolic (15 mmHg) drop in blood pressure or symptomatic presyncope occurred
14. Subject has a clinically significant unstable illness, for example hepatic impairment or renal insufficiency, or cardiovascular, pulmonary, gastrointestinal, endocrine, rheumatological, immunological, infection, skin and subcutaneous tissue disorder or metabolic disturbance
15. Subject has a history of HIV infection
16. Subject has a history of marijuana abuse or dependence (except topical CBD) within 1 year of the screening visit
17. Subject has a history of alcohol, drug abuse or dependence (except nicotine dependence) within 2 years of the screening visit
18. Subject has a history of cancer within 5 years of the screening visit (other than non-melanoma skin cancer, stable non-progressive prostate cancer not requiring treatment or in situ cervical cancer)
19. Subject has any surgical or medical condition which may significantly alter the absorption of any drug substance including, but not limited to, any of the following:

    1. History of major gastrointestinal tract surgery (e.g. bariatric surgery)
    2. Currently active inflammatory bowel syndrome
20. Female subject who is pregnant, nursing or of childbearing potential and not practicing effective contraception
21. Subject is required to take excluded medications as specified in the Excluded Medications section below.
22. Subject has a known or suspected intolerance or hypersensitivity to the study drug, closely related compounds, or any of their stated ingredients
23. Subject resides in hospital or moderate to high dependency continuous care facility
24. Evidence of clinically relevant pathology that in the investigator's opinion could interfere with the study results or put the subject's safety at risk

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2026-10-26 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to end of treatment in ADAS-Cog13 and ADCS-iADL | 78 weeks
  Primary Efficacy Endpoint
  • Co-primary endpoints of Alzheimer's Disease Assessment Scale cognitive subscale, 13-items (ADAS-Cog13) with a score range of 0-85 (higher scores indicating greater dysfunction) and Alzheimer's Disease Cooperative Study Instrumental Activities of Daily Living (ADCS-iADL) with a score range of 0-56 (lower scores indicating worse performance), in subjects with a clinical diagnosis of mild-to-moderate AD and biological diagnosis of AD pathology. ADAS-cog 13

SECONDARY OUTCOMES:
Change from Baseline to End of Treatment in plasma AB42/40 ratio, in subjects with a clinical diagnosis of mild-to-moderate AD and biological diagnosis of AD pathology | 78 weeks
Change from Baseline to End of Treatment in disease stage progression on the Clinical Dementia Rating Scale-Global (CDR-Global), in subjects with a clinical diagnosis of mild-to-moderate AD and biological diagnosis of AD pathology | 78 weeks
  CDR global score has a range of 0-3 with a higher score indicating greater dementia severity
Change from baseline to end of treatment in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB), in subjects with a clinical diagnosis of mild-to-moderate AD and biological diagnosis of AD pathology | 78 weeks
  CDR-SB has a score range of 0-18 with a higher number indicating greater dementia severity
Change from Baseline to End of Treatment on the integrated Alzheimer's Disease Rating Scale (iADRS), in subjects with a clinical diagnosis of mild-to-moderate AD and biological diagnosis of AD pathology | 78 weeks
  The iADRS is a composite scale that is calculated as a linear combination of total scores of the two individual components, the ADAS-Cog13 (score range 0-85) and the instrumental items of the ADCS-ADL (ADCS-iADL; score range 0-56)1 • The iADRS score ranges from 0-141 with lower scores indicating worse performance.

OTHER OUTCOMES:
Additional Endpoints (Exploratory) • Change from Baseline to End of Treatment in plasma proteomic biomarker levels (i.e. Neurogranin, GFAP, MTBR-243) | 78 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Didsbury, Chief Executive Officer, Ph.D, Study Director — T3D Therapeutics, Inc.
Locations (1):
- T3D Therapeutics, Inc., Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided